CLINICAL TRIAL: NCT06934837
Title: Evaluation of Swallowing Muscles Using Ultrasonography and Shear Wave Elastography in Patients Receiving Radiotherapy for Nasopharyngeal Carcinoma Diagnosis
Status: Completed | Type: Observational
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Collaborators: Selcuk University (Other)
Responsible Party: Principal Investigator, Fatih İkiz, Principal Investigator, Konya Beyhekim Training and Research Hospital
Other Study IDs: SUFM
Record Dates: First submitted 2025-04-06; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Patients Receiving Radiotherapy for Nasopharyngeal Carcinoma Diagnosis; Ultrasonography and Shear Wave Elastography; Evaluation of Swallowing Muscles
Keywords: Dysphagia; Nasopharynx cancer; SWE; Swallowing disorders
MeSH Terms: conditions — Deglutition Disorders; Nasopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Nasopharynx canser (disease group): 16 Stage I nasopharynx cancer patients receiving radiotherapy
- Control (healthy) group: 16 healthy volunteers from the otorhinolaryngology outpatient clinic

SUMMARY:
The aim of this study is to evaluate the mylohyoid, geniohyoid and digastric muscles in patients with radiotherapy-induced dysphagia due to nasopharynx cancer using ultrasonography and shear wave elastography (SWE).

DETAILED DESCRIPTION:
Post-radiotherapy swallowing dysfunction evaluation was carried out using fibreoptic endoscopic evaluation (FEES), ultrasonography of the swallowing muscles, shear wave elastography and swallowing assessment scale between the dates of 01/01/2023 and 01/06/2023.

All patients were interviewed to obtain detailed medical histories. Following this, standardized swallowing assessments were administered, including the Eating Assessment Tool (EAT-10) and the M.D. Anderson Dysphagia Inventory (MDADI). Head and neck examination, endoscopic examination and fibreoptic endoscopic swallowing assessment were performed at the Otorhinolaryngology, Head and Neck Surgery clinic. Penetration Aspiration Score (PAS) was determined by the experienced faculty member. Afterwards, an experienced radiologist performed neck ultrasonography and shear wave elastography (SWE) using an Aplio 500 Platinium Ultrasonography system (Toshiba Medical Systems, Japan) equipped with high-frequency linear transducer (frequency range = 5-14 MHz). With SWE, the stiffness values of the mylohyoid, geniohyoid and digastric muscles were measured in m/s and kPa, and their thickness was measured in mm. The tissue elasticity was outlined using a colour-coded system ranging from dark blue indicating least stiffness to red representing greatest stiffness, with a default measurement range of 0-120 kPa. The elastic value E (kPa) is calculated using the equation E = 3 ρ (m/s) 2. In the equation, m/s represents the shear wave propagation speed, and ρ represents the tissue density (approximately 1 in humans). All patients receiving radiotherapy were treated in our hospital's radiation oncology clinic for Stage I nasopharyngeal cancer received 70 Gy (2,12 Gy/Gun) gross tumour value (CTV70), with 5-10 mm margin for microscopic spread, delivered according to the International Commission on Radiation Units and Measurements (ICRU) Reports 50 and 62 guidelines. After obtaining the data, comparisons between the groups and correlations between the quantitative data were assessed using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria

Patient Group:

* Volunteered for the study.
* Aged 18-65 years.
* Diagnosed with Stage I nasopharynx cancer.
* Completed radiotherapy treatment at least 12 months prior to the study.
* No additional cancer diagnoses.
* No history of chemo-radiotherapy.
* No prior head-neck trauma or surgery.
* No rheumatologic or neuromuscular disorders.
* No pre-existing swallowing disorders.
* Control Group (Healthy Volunteers):

Control group:

* Aged 18-65 years.
* No history of head and neck cancer.
* No prior neck surgery or trauma.
* No radiotherapy to the head and neck region.
* No rheumatologic or neuromuscular disorders.
* No central haemorrhagic or ischemic disease.
* No pre-existing swallowing disorders.

Exclusion Criterias:

* Younger than 18 years or older than 65 years.
* Any history of neck interventions (e.g., for cancer metastasis, cervical spine surgery, trauma).
* Presence of systemic conditions potentially causing dysphagia (e.g., neurological, rheumatological, metabolic, or muscular disorders).
* Previous radiotherapy for reasons other than Stage I nasopharynx cancer (in the patient group).
* Any other cancer diagnosis besides Stage I nasopharynx cancer (in the patient group).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 or older than 65 years receiving radiotherapy, presented with dysphagia.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Swallowing muscle thickness | 12 months after radiotherapy.
  Right and left digastric - mylohyoid muscle thickness, as well as geniohyoid thickness using ultrasonography and Shear Wave Elastography. The thickness values of the mylohyoid, geniohyoid and digastric muscles were measured in mm by experienced radiologist.
Swallowing muscle pressure | 12 months after radiotherapy.
  Right and left digastric - mylohyoid muscle pressure, as well as geniohyoid pressure using ultrasonography and Shear Wave Elastography. The outcome pressure is measured in kPA by an experienced radiologist .
Swallowing muscle velocity | 12 months after radiotherapy.
  Right and left digastric - mylohyoid muscle velocity, as well as geniohyoid velocity using ultrasonography and Shear Wave Elastography. The velocity values of the mylohyoid, geniohyoid and digastric muscles were measured in m/s by an experienced radiologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Selçuk University Faculty of Medicine Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All data generated or analysed during this study are included in this research. Further inquiries or requests regarding the patient data can be directed to the corresponding author when necessary.